CLINICAL TRIAL: NCT04354909
Title: Soluble CD95 Ligand Role in the Pathophysiology of Non-infectious Active Uveitis
Acronym: UVE-FAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/43
Record Dates: First submitted 2020-03-16; First posted 2020-04-21 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Non-Infectious Active Uveitis
Keywords: Non infectious active uveitis; Soluble-CD95-Ligand

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biological samples: levels of s-CD95-L (ELISA test)
  Interventions: Other: s-CD95-L

INTERVENTIONS:
Other: s-CD95-L — levels of s-CD95-L (ELISA test)

SUMMARY:
The study aims at defining the role of soluble CD95 Ligand in the physiopathology of the non-infectious uveitis. Soluble CD95 Ligand might have a prognostic interest as well as potential for the discovery of new therapeutic strategies

DETAILED DESCRIPTION:
Non-Infectious active uveitis is a severe inflammatory ocular disease which can expose to the blindness. Actually, the knowledge of the physiopathology of uveitis stay poorly. CD95 Ligand (CD95-L) belongs to a TNF (tumor necrosis factors) receptor family. It knows to play a preponderant role to maintain the eye immune privilege. In particular conditions depending on immunologic environment, CD95-L has pro-inflammatory properties and can interact with Th17 lymphocytes and neutrophils, two cells implicated in non-infectious uveitis. The hypothesis is that s-CD95-L levels might be a prognostic factor in non-infectious uveitis and the study of the molecular mechanisms involved could provide new therapeutic targets.

This study will recruit 100 patients with non-infectious uveitis followed in Bordeaux University Hospital. Among classical disease activity information, blood samples will be collected during to assess s-CD95-L. Fundamental research will be realized on patients' sample to evaluate underlying molecular mechanisms.

Clinical and biological disease activity, treatment and outcomes will be studied in correlation with s-CD95-L to describe their potential prognostic role. Patients will be followed at regular intervals, accordingly to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-infectious uveitis according to the SUN (Standardization of the Uveitis Nomenclature) working Group;
* Age ≥ 18 years;
* being affiliated to health insurance,
* willing to participate.

Exclusion Criteria:

* Pregnant or breastfeeding women,
* patient under legal protection measure ,
* poor understanding of the French language

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with non-infectious uveitis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
levels of s-CD95-L | Baseline
  levels of s-CD95-L (ELISA test) in sera of non-infectious uveitis patients

SECONDARY OUTCOMES:
Correlation between levels of s-CD95-L and Disease activity score | Baseline, Month 3
  Correlation between levels of s-CD95-L and Disease activity score (as defined by ophthalmologic examination)
Th17 dosage | Baseline, Month 3
  Th17 dosage
polynuclear neutrophils levels | Baseline, Month 3
  polynuclear neutrophils levels (Flow cytometry)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No